CLINICAL TRIAL: NCT05437640
Title: Optimizing Protein Patterns for Skeletal Muscle Preservation and Sleep in the Medical Management of Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Christine Ferguson, PhD, RD, LD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300009538; P30DK056336 (NIH)
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Diet; Protein; Skeletal Muscle; Sleep
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: PD participants randomly assigned to first adhere to either the Protein Consistent Diet or Protein Redistribution Diet for 2 weeks. Participants will enter a 1-week washout period between the diets where they follow their typical diet and then follow the other diet prescription for 2 weeks.
Who Masked: Outcomes Assessor
Masking Description: Interpretation of blood biomarkers will be blinded to the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein Redistribution Diet (Active Comparator): PD participants may first be randomized to follow the Protein Redistribution Diet followed by the Protein Consistent Diet.
  Interventions: Behavioral: Protein Redistribution Diet
- Protein Consistent Diet (Active Comparator): PD participants may first be randomized to follow the Protein Consistent Diet followed by the Protein Redistribution Diet.
  Interventions: Behavioral: Protein Consistent Diet

INTERVENTIONS:
Behavioral: Protein Redistribution Diet — PD participants will be instructed by a Registered Dietitian to consume 10 grams or less of protein until their evening meal. They will then consume a high protein evening meal to meet their protein needs. They will receive one-on-one education and supportive materials to follow diet plan.
  Other Names: PRD
  Arms: Protein Redistribution Diet
Behavioral: Protein Consistent Diet — PD participants will be instructed by a Registered Dietitian to consume 20-30 grams of protein per meal. They will receive one-on-one education and supportive materials to follow diet plan.
  Other Names: PCD
  Arms: Protein Consistent Diet

SUMMARY:
The purpose of this pilot study is to generate preliminary data on the impact of the dietary protein pattern on markers of skeletal muscle health and drug efficacy in Parkinson disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a complex neurological disease that affects ~6.1 million people worldwide - mostly older adults >60 years. The most effective treatment for PD is dopaminergic therapy, particularly levodopa (Ldopa). People with PD have variable responses to Ldopa, including degrees of motor fluctuations (MF) throughout the day. The half-life of Ldopa is ~1.5 h and therefore, dosage and timing are essential to mitigate MF. Ldopa is a large neutral amino acid (LNAA), and the bioavailability of Ldopa is compromised when simultaneously ingested with LNAA (e.g., leucine). Both Ldopa and LNAAs from food are absorbed through the same intestinal transporter, but LNAAs from food are preferentially absorbed by the enterocyte, limiting the bioavailability of Ldopa. Thus, the scientific community often recommends the protein-redistribution diet (PRD). With PRD, patients limit protein (<10 g) at the desired time of medication efficacy (daytime) and meet their protein needs during the evening meal (~70+g). There are deleterious implications of the PRD for older adults with PD; consumption of >30 g of protein, in a single meal, will not sufficiently increase muscle protein synthesis. Additionally, the impact of the PRD on skeletal muscle quality and function has not been determined, and it is unclear, based on prior studies, whether the PRD enhanced drug absorption. Therefore, the objective of this study is to address these gaps in knowledge. This study will quantify the effects of dietary protein pattern on skeletal muscle in PD; determine the effects of dietary protein pattern on sleep quality in PD. This study is an acute, 5-week, crossover intervention with PD participants randomly assigned to first adhere to either the PCD or PRD. Participants will receive diet prescriptions and meal plans for their respective diet, and outcome measures will be assessed at days 0, 14, 21, and 35.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic PD for 5 or more years
* 45 years or older
* On a stable levodopa regimen for 3 or more months
* Self-reported to experience motor fluctuations

Exclusion Criteria:

* Following a specific diet that would preclude participation
* Renal disease
* Deep brain stimulation
* Known narcolepsy
* Untreated sleep apnea
* Any condition that, in the opinion of the investigator, will preclude the participant from successfully or safely completing study procedures

Ages: 45 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine C Ferguson, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Protein Consistent Diet, Then Protein Redistribution Diet: PD participants first were randomized to follow the Protein Consistent Diet for 2 weeks. After a washout period of 2 weeks, they then followed by a Protein Redistribution Diet.
- Protein Redistribution Diet, Then Protein Consistent Diet: PD participants first were randomized to follow a Protein Redistribution diet. After a washout period of 2 weeks, they then followed a Protein Consistent Diet.
Period: First Intervention (2 Weeks)
Arm/Group | Protein Consistent Diet, Then Protein Redistribution Diet | Protein Redistribution Diet, Then Protein Consistent Diet
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Protein Consistent Diet, Then Protein Redistribution Diet | Protein Redistribution Diet, Then Protein Consistent Diet
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Protein Consistent Diet, Then Protein Redistribution Diet | Protein Redistribution Diet, Then Protein Consistent Diet
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Participants: All participants were scheduled to follow both dietary interventions. One participant withdrew during the washout phase. Enrolled n=12, final n=11
Arm/Group | Total Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 65 [55 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Markers of Skeletal Muscle Metabolism GDF15
Description: Serum Growth Differentiation Factor 15 (GDF15)
Time Frame: Baseline to 5 weeks
Reporting Status: Not Posted, anticipated posting 2025-06

2. Primary Outcome: Change in Markers of Skeletal Muscle Metabolism FGF21
Description: Serum Fibroblast Growth Factor 21 (FGF21)
Time Frame: Baseline to 5 weeks
Reporting Status: Not Posted, anticipated posting 2025-06

3. Primary Outcome: Change in Handgrip Strength
Description: Handgrip strength assessed via digital dynamometer
Time Frame: Baseline to 5 weeks
Reporting Status: Not Posted, anticipated posting 2025-06

4. Primary Outcome: Change in Sleep Efficiency
Description: Sleep efficiency assessed via actigraphy
Time Frame: Baseline to 5 weeks
Reporting Status: Not Posted, anticipated posting 2025-06

5. Primary Outcome: Change in Motor Symptoms
Description: Motor symptoms assessed via the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II. Part II ranges from 0-52 with higher scores indicating greater symptom severity.
Time Frame: Baseline to 5 weeks
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Protein Redistribution Diet | Protein Consistent Diet
Number analyzed (Participants) | 11 | 12
Score
  Baseline | 11.27 (5.57) | 9.58 (7.75)
  Post-Diet | 9.45 (5.97) | 9.42 (4.94)

6. Secondary Outcome: Change in Physical Activity
Description: Physical activity assessed via actigraphy
Time Frame: Baseline to 5 weeks
Reporting Status: Not Posted, anticipated posting 2025-06

7. Secondary Outcome: Change in Total Parkinson Symptoms
Description: Parkinson-related symptoms assessed by total MDS-UPDRS score
Time Frame: Baseline to 5 weeks. Total score ranges from 0-260 with higher scores indicating greater symptom severity.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Protein Redistribution Diet | Protein Consistent Diet
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 52.09 (20.92) | 51.17 (21.04)
  Post-Diet | 47.18 (19.15) | 48.75 (20.52)

ADVERSE EVENTS:
Time Frame: Adverse event information was assessed during the study period (5 weeks)
Groups:
- Protein Consistent Diet: PD participants will be instructed by a Registered Dietitian to consume 20-30 grams of protein per meal. They will receive one-on-one education and supportive materials to follow diet plan.
  One participant withdrew during the washout phase after completing the Protein Consistent Diet.
- Protein Redistribution Diet: PD participants will be instructed by a Registered Dietitian to consume 10 grams or less of protein until their evening meal. They will then consume a high protein evening meal to meet their protein needs. They will receive one-on-one education and supportive materials to follow diet plan.
  No participants experienced adverse events in PRD phase.
Arm/Group | Protein Consistent Diet | Protein Redistribution Diet
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protein Consistent Diet (N=12) | Protein Redistribution Diet (N=12)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Migraines (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT05437640/Prot_SAP_000.pdf